CLINICAL TRIAL: NCT05125276
Title: Less Bleeding by Omitting Aspirin in Non-ST-segment Elevation Acute Coronary Syndrome Patients
Acronym: LEGACY
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, J.P.S Henriques, Prof. Dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL79129.018.21
Record Dates: First submitted 2021-11-08; First posted 2021-11-18 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Non ST Segment Elevation Acute Coronary Syndrome
MeSH Terms: interventions — N-acetyl-S-(alpha-methyl-4-(2-methylpropyl)benzeneacetyl)cysteine 4-(nitrooxy)butyl ester; Aspirin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional arm (Experimental): No aspirin
  Interventions: Drug: No aspirin
- Control arm (Active Comparator): Aspirin (75-100 mg once daily)
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: No aspirin — No aspirin
  Arms: Interventional arm
Drug: Aspirin — 75-100 mg once daily
  Arms: Control arm

SUMMARY:
Rationale: Dual antiplatelet therapy, consisting of aspirin and a P2Y12-inhibitor, reduces the risk of stent thrombosis, myocardial infarction and stroke after coronary stent implantation. Inevitably, it is also associated with a higher risk of (major) bleeding. Given the advances in stent properties, stenting implantation technique and pharmacology, it may be possible to treat patients with a single antiplatelet strategy by completely omitting aspirin.

Objective: This study will assess whether omitting aspirin reduces the rate of major or minor bleeding while remaining non-inferior to the current standard of care with regards to ischemic events in patients with non-ST segment elevation acute coronary syndrome.

Study design: Open-label, multicentre randomized controlled trial.

Study population: Adult patients presenting with non-ST segment elevation acute coronary syndrome undergoing percutaneous coronary intervention.

Intervention: In the intervention group aspirin will be completely omitted from the antiplatelet regimen in the 12 months following PCI.

Main study endpoints: The primary bleeding endpoint is major or minor bleeding defined as Bleeding Academic Research Consortium type 2, 3 or 5 bleeding at 12 months. The primary ischemic endpoint is ischemic events defined as the composite of all-cause death, myocardial infarction and stroke at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of NSTE-ACS (i.e. NSTEMI or unstable angina)
* Successful PCI (according to the treating physician)

Exclusion Criteria:

* Known allergy or contraindication for aspirin or all commercially available P2Y12-inhibitors (i.e. ticagrelor, prasugrel and clopidogrel)
* Concurrent use of oral anticoagulants (e.g. because of atrial fibrillation)
* Ongoing indication for DAPT at admission (e.g. due to recent PCI or ACS)
* Planned surgical intervention within 12 months of PCI
* Pregnant or breastfeeding women at time of enrolment
* Participation in another trial with an investigational drug or device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3090 (Estimated)
Dates: Start 2022-05-13 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Bleeding endpoint | 12 months
  The primary bleeding endpoint at 12 months is major or minor bleeding defined as BARC type 2, 3 or 5 bleeding
Ischemic endpoint | 12 months
  The primary ischemic endpoint at 12 months is the composite of all-cause mortality, myocardial infarction and stroke

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Amsterdam UMC, location AMC, Amsterdam
  - Amsterdam UMC, location VUmc, Amsterdam

IPD SHARING:
Plan to Share IPD: Undecided